CLINICAL TRIAL: NCT00887601
Title: A 4-Period, Placebo-Controlled, Crossover Study to Evaluate the Utility and Feasibility of BOLD fMRI and Cerebral Blood Flow Measurements as Biomarkers for Cognition Enhancing Drugs (Donepezil and MK3134)
Brief Title: BOLD Functional Magnetic Resonance Imaging (fMRI) and Cerebral Blood Flow Measurements as Biomarkers for Cognition Enhancing Drugs (3134-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3134-006; 2009_583
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part I (Experimental): Subjects will receive placebo, MK3134, and donepezil in one of four treatment sequences.
  Interventions: Drug: MK3134; Drug: Comparator: Placebo; Drug: Donepezil
- Part II (Experimental): Subjects will receive placebo and three different doses of MK3134 (1 mg, 5 mg, and 25 mg) in one of four treatment sequences.
  Interventions: Drug: Comparator: Placebo; Drug: MK3134

INTERVENTIONS:
Drug: MK3134 — Single dose 25 mg (5 x 5 mg) MK3134 capsules in one of the four treatment periods.
  Arms: Part I
Drug: Comparator: Placebo — Placebo capsules only in one of the four treatment periods.
Drug: Donepezil — Single dose 5 mg donepezil capsules in two of the four treatment periods.
  Other Names: Aricept
  Arms: Part I
Drug: MK3134 — Single doses of 1 mg, 5 mg, or 25 mg MK3134 capsules in the assigned treatment periods
  Arms: Part II

SUMMARY:
This study will evaluate functional magnetic resonance imaging (fMRI) and methods for measuring drug induced changes in cerebral blood flow as biomarkers for attention-improving drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a nonsmoker
* Subject is in generally good health
* Subject has normal (or corrected to normal) vision and hearing
* Subject is right-handed

Exclusion Criteria:

* Subject has a history of any illness that would make participation unsafe or would make the study results difficult to interpret
* Subject has a history of stroke, seizures, or major neurological disorders
* Subject has a history of cancer
* Subject has permanent cosmetic or metallic implants that would interfere with measurements
* Subject has a history of sleep apnea
* Subject has a history of head injury/trauma

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Part I: Difference in number of voxels showing a positive response after treatment with donepezil and placebo | 3.5 to 4.5 hours after study drug administration
Part I: Difference in number of voxels activated for both faces and scenes after treatment with donepezil and placebo | 3.5 to 4.5 hours after study drug administration
Part II: Number of voxels showing a positive response after varying doses of MK3134 compared to placebo | 3.5 to 4.5 hours after study drug administration
Part II: Number of voxels activated for both faces and scenes after varying doses of MK3134 compared to placebo | 3.5 to 4.5 hours after study drug administration

SECONDARY OUTCOMES:
Part I: Difference in arterial transit time as measured by arterial spin labeling after treatment with donepezil and placebo | 3.5 to 4.5 hours after study drug administration
Part I: Difference in Pulsatility index after treatment with donepezil and placebo | 5 hours after study drug administration
Part I: Test-retest reproducibility of the BOLD fMRI and cerebral blood flow measurements in donepezil treated subjects | 1 to 5 weeks
Part II: Change in arterial transit time after treatment with placebo and varying doses of MK3134 | 3.5 to 4.5 hours after study drug administration
Part II: Change in Pulsatility index after treatment with placebo and varying doses of MK3134 | 5 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC